CLINICAL TRIAL: NCT07125248
Title: Outcomes of Transhiatal Drain Placement in Esophagectomy, a Randomised Control Trial
Brief Title: Outcomes of a Single Chest Drain vs Two Drains
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Dr Saeed Sarwar, Doctor, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 190/DME/KM
Record Dates: First submitted 2025-08-04; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pleura; Effusion; Esophageal Adenocarcinoma; Esophageal Anastomotic Leak
MeSH Terms: conditions — Pleural Effusion; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral chest drains group (Experimental): Participants in this group will have bilateral intercostal chest tubes placed during surgery.
  Interventions: Procedure: Bilateral chest tube placement
- Single drain group (Experimental): Paricipants in this group will have a single transhiatal drain placed in mediastinum that would be brought out through abdomen
  Interventions: Procedure: Single drain placement

INTERVENTIONS:
Procedure: Bilateral chest tube placement — Bilateral chest tubes will be passed in this intervention group through intercostal spaces
  Arms: Bilateral chest drains group
Procedure: Single drain placement — A single transhiatal drain will be placed in mediastinum in this group
  Arms: Single drain group

SUMMARY:
Esophagectomy is a major surgical procedure done for carcinoma of esophagus. Usually bilateral chest tubes are placed in surgery for prevention of fluid accumulation in chest. However such procedure limits patients mobility and increases severity of pain. recent studies suggest that a single drain can be safe and effective. our study aims to compare the results of two chest tubes vs one.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing open esophagectomy for carcinoma of esophagus

Exclusion Criteria:

* Non consenting individuals esophagectomy for benign disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Chest expansion | On postoperative day 1 and day 3 .
  Chest expansion will be observed by chest xray postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber teaching hospital, Peshawar, Khyberpukhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patients data will be confidential